CLINICAL TRIAL: NCT05260957
Title: ML43165 - Single Arm Phase 2 Trial of an FDA Approved Anti-CD19 CAR-T Therapy Followed by Mosunetuzumab and Polatuzumab Consolidation for the Treatment of Refractory/Relapsed Aggressive NHL.
Brief Title: CAR-T Cell Therapy, Mosunetuzumab and Polatuzumab for Treatment of Refractory/Relapsed Aggressive Non-Hodgkin's Lymphoma (NHL).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lazaros Lekakis (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lazaros Lekakis, Associate Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210828
Record Dates: First submitted 2022-02-15; First posted 2022-03-02 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Refractory Non-Hodgkin Lymphoma; Relapsed Non Hodgkin Lymphoma; Aggressive Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — polatuzumab vedotin; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination CAR-T Cell Therapy, Mosunetuzumab + Polatuzumab (Experimental): Participants will receive study treatment in three phases: Induction Phase, CAR-T Treatment Phase and Consolidation Phase.
  During the Induction Phase (Days -42, through -6), participants will receive Mosunetuzumab on Days -42, -35, -28, and -7; and Polatuzumab on Day -28. On Day -6, participants will be evaluated in clinic.
  During the CAR-T Treatment Phase (Days -5, through Day 0), participants will receive lymphodepleting chemotherapy for three consecutive days beginning on Day -5, followed by CAR-T Cell therapy via infusion on Day 0.
  During the Consolidation Phase (Days +1 through +90), participants will receive Mosunetuzumab on Day +14; and combination Mosunetuzumab and Polatuzumab on Days +35, +56 and +77.
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab; Biological: CAR-T Cell Therapy

INTERVENTIONS:
Drug: Mosunetuzumab — Induction Phase (Days -42 through -7):
  * 1 mg of Mosunetuzumab administered via intravenous (IV) infusion (given as per treatment guidelines) on Day -42.
  * 2 mg of Mosunetuzumab administered via intravenous (IV) infusion (given as per treatment guidelines) on Day -35.
  * 60 mg of Mosunetuzumab administered via intravenous (IV) infusion on (given as per treatment guidelines) on Days -28 and -7.
  Consolidation Phase (Day +1 through Day +90): 30 mg IV Mosunetuzumab administered via intravenous (IV) infusion (given as per treatment guidelines) on Days +14, +35, +56 and +77.
  Other Names: BTCT4465A
Drug: Polatuzumab — Induction Phase (Days -42 through -7): 1.8mg/kg of Polatuzumab administered via intravenous (IV) infusion (given as per treatment guidelines) on Day -28.
  Consolidation Phase (Days +1 through +90): 1.8mg/kg of Polatuzumab administered via intravenous (IV) infusion (given as per treatment guidelines) on Days +35, +56 and +77.
  Other Names: Polatuzumab Vedotin; RO5541077; Polivy
Biological: CAR-T Cell Therapy — Participants will receive CAR-T Cell therapy via infusion on Day 0 (given as per treatment guidelines). Prior to CAR-T Cell Therapy, participants will begin receiving lymphodepleting chemotherapy on Days -5 through -3 (given as per treatment guidelines).
  Other Names: Chimeric antigen receptor T-Cell Therapy

SUMMARY:
The purpose of this research study is to test if a combination treatment of chimeric antigen receptor (CAR) T-cell therapy, Mosunetuzumab, and Polatuzumab Vedotin will result in tumor reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of:

   1. Diffuse large B cell lymphoma (DLBCL) not otherwise specified. Patients with primary cutaneous DLBCL of leg-type are eligible if the lymphoma expresses cluster of differentiation 19 (CD19) and if the insurance approves the CAR-T therapy. Similarly. Large cell transformation of nodal or extra-nodal marginal zone lymphoma is eligible only if the insurance allows and the disease shows strong CD19 positivity. On the other hand, post-transplant lymphoproliferative disorders (PTLD) are not allowed due to the frequently required continuation of immunosuppression to avoid organ rejection.
   2. Primary mediastinal B cell lymphoma (PMBCL)
   3. Transformed follicular lymphoma (TFL). An untransformed follicular lymphoma grade 3B will be considered on a case by case basis, since the genetic signature of grade 3B follicular lymphoma frequently resemble that of DLBCL and the large lymphomatous cells just happen to be organized in a follicular pattern. Recently, Breyanzi has an FDA indication for follicular lymphoma grade 3B.
   4. High grade B cell lymphoma (HGBL), other than B-lymphoblastic lymphoma
   5. Mantle Cell lymphoma (MCL)
   6. Burkitt lymphoma (BL): Although very few reports inform us about the outcome of relapsed/refractory BL, encouraging activity including CRs have been reported with CAR-T and these patients are in need because they do not have enough options available. We will need insurance approval for such enrollment.
2. Additionally, the lymphoma has to be in one of the following status:

   1. Primary refractory which for the purpose of this study is defined as failure to obtain any response (PR or CR) after at least 3 cycles of anthracycline-based therapy or persistent disease after 6 cycles of anthracycline-based therapy as documented by a PET/CT scan that is done no later than 2 months after the last (usually the 6th) cycle of primary chemotherapy. In questionable cases, a biopsy should confirm persistence of disease as part of standard of care. In case of mantle cell lymphoma, the primary therapy if does not include an anthracycline, should include either high doses of cytarabine +/-bendamustine and an anti-CD20 antibody (usually rituximab).
   2. Relapsed disease that fails to respond (CR or PR) after at least 2 cycles of a platinum and/or cytarabine-based chemotherapy. For the purpose of this study, appropriate regimens include: rituximab, ifosfamide, carboplatin and etoposide (R-ICE), rituximab, dexamethasone, cytarabine, and cisplatin (R-DHAP), rituximab dexamethasone cytarabine oxaliplatin (R-DHAOx), rituximab, gemcitabine, cisplatin, and dexamethasone (R-GDP). Rituximab, gemcitabine, and oxaliplatin (R-Gem-Ox) is considered appropriate if the patient fails to obtain at least a PR after 4 doses of oxaliplatin. Patients with MCL who relapse after an anthracycline, bendamustine or cytarabine-based regimen, should have failed two salvage attempts: a molecularly targeting-based regimen including at least a Bruton's tyrosine kinase (BTK) inhibitor with or without venetoclax and a cytotoxic traditional second salvage regimen, unless the two salvage approaches are combined. For example if they fail a salvage with R-ICE + a BTK-inhibitor in combination, they are eligible without the need to be exposed to more therapy. Patients with PMBCL, they should also have failed a traditional salvage regimen and a programmed cell death protein 1 (PD-1) inhibitor-based salvage.
   3. Relapse after an autologous stem cell transplantation. At least 3 months should have lapsed between autologous stem cell infusion and initiation of pre-CAR-T lymphodepleting chemotherapy due to the risk of prolonged cytopenias.
3. At least one of the lymphoma lesions should be measurable. For the purpose of this study an involved nodal lesion should be at least 1.5 cm in the longest diameter, while extra-nodal lymphoma lesions should have their longest diameter ≥1.0 cm
4. Lymphoma cells need to be CD19 positive. In case of previous therapy with an anti-CD19 agent (including but not limited to blinatumomab, tafasitamab, loncastuximab tesirine), a new biopsy should be performed to confirm CD19 positivity.
5. The performance status of the patient as measured by the Eastern Cooperative Oncology Group (ECOG) performance scale should be 0 - 2 (ECOG performance status (PS):0-2).
6. Only adult patients will be eligible (patient age >18 years old). Patients up to 80 years old will be considered to participate in the study assuming they fulfill all the other inclusion criteria
7. The creatinine clearance as measured by the Cockcroft-Gault equation should be 50 mL/min or better (CrCl ≥ 50 mL/min).
8. Unless the patient has a known Gilbert syndrome, the total Bilirubin should be less that 1.5 x upper limit of normal (ULN) and both the transaminases (ALT and AST) should be less than 2.5 x ULN. The only exception to this rule is lymphoma infiltration of the liver where values of total Bilirubin up to 3 x ULN and transaminases up to 5 x ULN will be allowed after communication with the Principal Investigator (P.I. or his/her designee)
9. The ejection fraction of the left ventricle as it is estimated on the Echocardiogram (preferably) or on the multigated acquisition (MUGA) scan should be at least 45% (LVEF ≥ 45%).
10. The oxygen saturation of oxyhemoglobin on room air as measured by pulse oximetry should be at least 94% (O2Sat ≥ 94%). If a technical problem (artifact) is suspected on pulse oximetry, arterial blood gases will be obtained for more accurate measurement.
11. On the day of screening and assuming there will be no other than the protocol therapy, the patient should have at least the following:

    1. Absolute neutrophil count >1000/microliter,
    2. Hg> 8 grams/ deciliter
    3. Absolute lymphocyte count >250/microliter
    4. Platelet count >75,000/microliter
12. Patient should not have a transfusion of packed red blood cells (PRBCs) or platelets or receive erythropoietin analogues thrombopoietin receptor agonist (Tpo-mimetic), granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) for at least 5 days before the official determination of eligibility takes place.
13. Patient should sign an informed consent and be willing to comply with the anticipated labs and clinic visits and should be willing to be hospitalized and undergo the required invasive procedures as directed by the treating Investigator.
14. Female subjects should have a negative serum pregnancy test, unless they confirm their menopausal status and/or have undergone previous hysterectomy and/or oophorectomy.
15. Both men and women with childbearing potential should agree to use effective contraception for the duration of the treatment and for at least 1 year after the last treatment since medications (e.g. cyclophosphamide) that will be used in the protocol can be harmful for the embryo.

Exclusion Criteria:

1. Patients with EBV+DLBCL, plasmablastic lymphoma, human herpesvirus-8 (HHV-8) related B cell lymphoproliferative disorders including primary effusion lymphoma, anaplastic lymphoma kinase (ALK)+ LBCL, intravascular large B cell lymphomas, DLBCL associated with chronic inflammation, lymphomatoid granulomatosis, primary DLBCL of the CNS and T cell histiocyte rich LBCL will not be allowed because of different biology, frequent lack of CD19, difficulty in interpreting toxicity (as in the case of primary central nervous system (CNS) lymphoma) or some preliminary discouraging results with CAR-T as in the case of T-cell, histiocyte-rich large B cell lymphoma and Richter transformation of chronic lymphocytic leukemia (CLL).
2. Primary CNS lymphoma or secondary CNS involvement by lymphoma.
3. Similarly, patients with conditions that increase the risk of CNS toxicity will be excluded. Such conditions include but not limited to

   1. active seizure disorder for which an antiepileptic is taken,
   2. demyelinating diseases like multiple sclerosis
   3. history of ischemic or hemorrhagic stroke in the last 2 years
   4. Neurodegenerative disorders like Alzheimer and Parkinson
   5. Cerebral edema or hydrocephalus of any cause
4. Invasive sarcoma or carcinoma in the last 3 years, except from localized basal or squamous cell carcinomas of the skin, or cervical carcinoma in situ. Localized Gleason <7, prostate-specific antigen (PSA)<10 prostatic adenocarcinoma T1-2N0M0 under active surveillance is allowed.
5. Myocardial infarction or unstable angina or coronary revascularization within 6 months of protocol enrollment is not allowed. Stable angina that requires nitrates for pain relief is not allowed either because of concerns of hypotension during the CRS period.
6. Systemic hypertension that is not controlled with maximum three antihypertensives to a level of <160/100 precludes enrollment.
7. Uncontrolled invasive infection, including fungal pneumonia, fungal sinusitis or fungal encephalitis are not allowed and should be resolved completely before enrollment. Cytomegalovirus (CMV) viremia>200 copies/microliter or EBV viremia > 1000 copies/microliter are not allowed unless treated completely in the case of CMV viremia and the patient then is placed on prophylactic letermovir.
8. Patients with history of macrophage activation syndrome (MAS)/hemophagocytic lymphohistiocytosis (HLH) and patients with known or suspected chronic active Epstein Barr Virus infection (CAEBV).
9. HIV positivity is allowed as long as the viral load of HIV-1 is less than 200 copies/microliter the last 3 months and the patient continue at least 3 antiretroviral agents during therapy.
10. Chronic hepatitis B should have been controlled to hepatitis B virus (HBV) viral load <200 copies/microliter and patients with chronic hepatitis B or even with just history of exposure to hepatitis B (hepatitis B core antibody positive but surface antigen negative) should be on suppressive therapy with entecavir, lamivudine or equivalent.
11. Patients with hepatitis C and clearance of the virus with previous therapy are allowed as long as they do not suffer from chronic liver dysfunction. Patients with chronic hepatitis C and normal hepatic function should be cleared by a Hepatologist before inclusion and at least an elastogram and an ultrasound should be performed to r/o well-compensated cirrhosis.
12. Autoimmune disorders including rheumatoid arthritis, severe psoriasis, systemic lupus erythematosus, scleroderma with pulmonary involvement, polymyositis, systemic vasculitis and inflammatory bowel disease requiring treatment with more than oral budesonide or nonacetylated salicylates are not allowed. Similarly pneumonitis, including cryptogenic organizing pneumonia, bronchiolitis obliterans or eosinophilic pneumonias or sarcoidosis affecting the lung parenchyma are not allowed. Guillain Barre, autoimmune hepatitis and autoimmune encephalitis as well as glomerulonephritis with nephrotic or nephritic syndrome are not allowed. Addison is allowed but prednisone daily dose should be less than 10 mg/d. Hashimoto thyroiditis is allowed as long as the patient has well controlled thyroid function with supplemental levothyroxine. Grave's disease has to be in excellent control with previous surgery or radioiodine or with methimazole with or without beta blockers but not glucocorticosteroids and patients will need endocrinology consultation before the enrollment.
13. Other causes of congenital or acquired immunodeficiencies other than common variable immunodeficiency or immunoglobulin A (IgA) deficiency are not allowed.
14. External drains including pericardial, pleural, peritoneal, external biliary drains or nephrostomies are not allowed.
15. Use of prednisone for any reason should not be >10 mg/d. All other systemic immunosuppressive agents are not allowed.
16. Any biologic agent interfering with the immune system function or cytotoxic chemotherapy are not allowed within 21 days of the first dose of mosunetuzumab. Radiation is not allowed within 14 days of the first mosunetuzumab administration. If temporary control of the lymphoma is required, only dexamethasone 20 mg/d for up to 5 days before the first administration of mosunetuzumab is allowed.
17. Patient should not have anti-human leukocyte antigen (HLA) antibodies that make them refractory to platelets transfusions.
18. If patients are on systemic antiplatelet or anticoagulant therapy, this therapy has to be stopped. Patients can continue low dose acetylsalicylic acid (ASA) up to 100 mg/d that will be also stopped when platelets drop below 75,000/microliter at any point during therapy. Non catheter-related deep venous thrombosis or pulmonary embolism that happened less than 3 months before protocol enrollment are not allowed.
19. Any cardiac disease in addition to left ventricular ejection fraction (LVEF) <45% that gives symptoms of heart failure (diastolic dysfunction or valvular abnormalities or dysrhythmias) and makes the patient belong to New York Heart Association (NYHA) II-IV functional group, automatically makes the patient ineligible.
20. Previous anti-CD19 CAR-T therapy is not allowed.
21. Uncontrolled Psychosis or cognitive impairment that makes the patient unable to make informed decisions preclude participation.
22. Previous solid organ transplantation precludes participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | 3 Months
  Complete Response (CR) rate will be reported as the percentage of participants achieving complete response (CR) to study treatment. Response to therapy will be assessed using Positron Emission Tomography (PET)/ Computerized Tomography (CT) scan following Lugano 2014 criteria (Cheson et al, Journal of Clinical Oncology (JCO), 2014) at 3 months (Day +90) of study treatment. For equivocal PET-CT results, biopsy will be performed after day +90 PET/CT to assess true CR or persistent lymphoma.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 months
  Overall response rate (ORR) will be reported as the percentage of participants achieving either complete response (CR) or partial response (ORR = CR + PR) to study treatment. Response to therapy will be assessed using Positron Emission Tomography (PET)/ Computerized Tomography (CT) scan following Lugano 2014 criteria (Cheson et al, Journal of Clinical Oncology (JCO), 2014) up to Day +90 of study treatment.
Progression free survival (PFS) Rate | Up to 2 years
  PFS is defined as the elapsed time from the date of starting treatment to the date of progression, or date of death from any cause; whichever comes first. PFS rate will be reported as the percentage of participants without progressive disease after start of treatment.
Overall Survival (OS) Rate | Up to 2 years
  Overall survival is defined as the elapsed time from the date of starting treatment to the date of death from any cause. OS rate will be reported as the percentage of participants still alive after start of treatment.
Minimal residual disease (MRD) negativity | Up to 1 year
  Minimal residual disease (MRD) negativity will be reported as the percentage of participants showing absence of measurable disease in peripheral blood after start of CAR-T Cell therapy. MRD negativity will be assessed by using the Clustering and Alignment of Polymorphic Sequences (CAPSeq) assay.
Duration of Response (DoR) | Up to 2 years
  Duration of response is defined as the elapsed time from date of complete response (CR) to the date of progression or death, whichever is first. DoR will be reported as the percentage of participants who relapsed after achieving CR on the Day +90 PET/CT scan. Relapse rate applies to unequivocal metabolic relapse or/and biopsy confirmed relapse among the patients who achieved CR on day +90 PET-CT
Toxicity Rate of CAR-T Cell Therapy: ICANS Events | Up to 6 months
  Toxicity rate of CAR-T Cell Therapy will be reported as the percentage of participants with treatment-emergent Immune Effector Cell Associated Neurotoxicity Syndrome (ICANS), after start of therapy, as evaluated by treating physician. The severity of ICANS events in participants will be assessed using American Society for Transplantation and Cellular Therapy (ASTCT) Consensus grading criteria (Lee et al, Biol Blood Marrow Transplant., 2019).
Toxicity Rate of CAR-T Cell Therapy: CRS Events | Up to 6 months
  Toxicity rate of CAR-T Cell Therapy will be reported as the percentage of participants with treatment-emergent Cytokine Release Syndrome (CRS) events, after start of therapy, as evaluated by treating physician. The severity of CRS events in participants will be assessed using American Society for Transplantation and Cellular Therapy (ASTCT) Consensus grading criteria (Lee et al, Biol Blood Marrow Transplant., 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Lazaros Lekakis, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No